CLINICAL TRIAL: NCT02835781
Title: Allogenic Acellular Dermal Matrix Use in Patients With Breast Reconstruction
Brief Title: Acellular Dermal Matrix in Breast Reconstruction
Acronym: Adermbrerec
Status: Completed | Type: Observational
Sponsor: University Hospital Bratislava (Other)
Collaborators: Comenius University (Other)
Responsible Party: Principal Investigator, Julius Hodosy, Principal investigator, University Hospital Bratislava
Other Study IDs: UHB/006/2015/MB
Record Dates: First submitted 2016-06-28; First posted 2016-07-18 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
Keywords: Breast Implants; Acellular Dermal Matrix
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammaplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Acellular dermal tissue after primary reconstruction will be harvested prior to second surgery with permanent implant.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acellular dermal matrix arm: The females undergoing breast reconstruction surgery after breast removal because of breast cancer. The breast reconstruction will be performed using acellular dermal matrix implantation.
  Interventions: Other: Acellular dermal matrix implantation

INTERVENTIONS:
Other: Acellular dermal matrix implantation — Acellular dermal matrix obtained from Central tissue bank, University Hospital Bratislava, will be used for acellular dermal matrix implantation.
  Other Names: breast reconstruction

SUMMARY:
Allogenic acellular dermal matrix has been used in burn injuries or abdominal walls reconstructions. However, it is solely used in breast reconstructions after breast carcinoma amputation. The efficacy of such allogenic dermal matrix can be advantageous when compared to current treatment options, however, this has to be proved.

DETAILED DESCRIPTION:
This is a prospective study, where patients undergoing breast reconstruction surgery using acellular dermal matrix (ADM) with expander use in first phase of reconstruction will be included. The permanent breast implants will be implanted approximately half year during second surgery. Acellular dermal matrix is a soft tissue graft that is formed by decellularization, however with intact extracellular dermal matrix. Such structure is able to re-create adequate skeleton for host cells with subsequent incorporation and revascularization. The safety and appropriateness of such ADM in breast reconstruction surgery will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* total one-side mastectomy due to breast cancer
* age between 18-60 years

Exclusion Criteria:

* failure to obtain signed informed consent

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The cohort will be selected from patients with breast cancer and in remission, sent to plastic and reconstruction surgery clinics for breast reconstruction after therapeutical mastectomy.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-01; Primary Completion 2014-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of complications in patients receiving acellular dermal matrix evaluated at 6 months after primary implantation | 6 months
  All patients between January 2010 and June 2014 undergoing primary ADM implantation will be evaluated at 6 months after implantation for early ex-plantations, inflammation, deformities of the implants, allergic reactions will be observed in patients undergoing primary ADM implantation at 6 months until second permanent implantation is performed.

SECONDARY OUTCOMES:
Histologic evaluation of ADM implants upon planned explantations | 6 months
  All patients between January 2012 and June 2014 after primary ADM transplantation will be evaluated. Analysis of cell composition, leukocytes at place, vessel formation and dysplasias will be performed
Satisfaction with breast reconstruction outcome evaluated by Breast-Q questionnaire | 2 years
  Physical and psychical as well as sexual well-being with outcome will be evaluated by specifically for this purpose developed questionnaire (The Breast-Q questionnaire) after permanent breast implant implantation at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Miroslav Bdzoch, MD, PhD, Study Director — University Hospital Bratislava, Pazitkova 4, Bratislava, Slovakia
Locations (1):
- University Hospital Bratislava, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bohac M, Varga I, Polak S, Dragunova J, Fedeles J Sr, Koller J. Delayed post mastectomy breast reconstructions with allogeneic acellular dermal matrix prepared by a new decellularizationmethod. Cell Tissue Bank. 2018 Mar;19(1):61-68. doi: 10.1007/s10561-017-9655-0. Epub 2017 Aug 16. PMID 28812172